CLINICAL TRIAL: NCT06183164
Title: The Effect of Awareness-Based Stress Reduction Program Applied to Breast Cancer Patients Receiving Chemotherapy on Symptom Management Psychological Resilience and Quality of Life
Brief Title: Awareness Based Stress Reduction Program Applied to Breast Cancer Patients Receiving Chemotherapy
Acronym: Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08/06/2023
Record Dates: First submitted 2023-11-30; First posted 2023-12-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Patients Receiving Chemotherapy
Keywords: life quality mindfulness psychological resilience symptom management

STUDY DESIGN:
Intervention Model Description: This study is an exprimental study with pre-test, intermediate test and post-test control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): The program lasts eight weeks, with face-to-face group meetings for 2-2.5 hours per week and applications requested from the patient. It is a program in which various mindfulness practices are used consecutively for eight weeks and completed with a six-hour silence (retreat) day at the end of the eight weeks.
  Interventions: Other: Mindfulness: Awareness-Based Stress Reduction Program
- Control group (No Intervention): Routine main tenance will be applied.

INTERVENTIONS:
Other: Mindfulness: Awareness-Based Stress Reduction Program — The mindfulness-based stress reduction program was applied to the patients in the experimental group once a week, for 150 minutes, for 8 weeks and 8 times in total. Then, an intermediate test is applied to the patients. After the interim test, patients are asked to repeat the mindfulness-based stress reduction program individually for 8 weeks (between weeks 8-16). In addition, after the conscious awareness-based stress reduction program is applied to the patients in the experimental group by the researcher, the 'Conscious Awareness-Based Stress Reduction Program' booklet prepared by the researcher is given to the patients as a guide. experimental group.
  Arms: Mindfulness

SUMMARY:
Implementation of awareness-based stress reduction program in breast cancer patients receiving chemotherapy and examining its effects on psychological resilience, symptom management and quality of life.

DETAILED DESCRIPTION:
The conscious awareness-based stress reduction program is a program that lasts eight weeks, each session lasting 2-2.5 hours and including a 6-hour silence day. In order to apply the mindfulness stress reduction program to the experimental group, the 'Conscious Awareness Stress Reduction Program day and time were determined for 30 breast cancer patients receiving chemotherapy who met the inclusion criteria and were sampled. It was applied to the patients in the experimental group, once a week for 150 minutes, lasting 8 weeks, and consisting of 8 times in total. Then, an intermediate test was applied to the patients. After the interim test, patients were asked to repeat the It applications individually for 8 weeks (between weeks 8-16). In addition, after It was applied to the patients in the experimental group by the researcher, the 'Conscious Awareness Stress Reduction Program booklet prepared by the researcher was given to the patients in order to provide a guide for the patients in the experimental group. During the implementation of the research, no intervention was applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Ability to communicate adequately
* No psychiatric problems
* Implementation of the Awareness-Based Stress Reduction Program is an obstacle
* Volunteering to participate in the research

Exclusion Criteria:

* Those who have communication problems
* Those with psychiatric problems
* Not agreeing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-29 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
ESTO SYMPTOM DIAGNOSIS SCALE | At the end of Sessions 16 ( each Session 1 days a week)
  The scale includes problems such as pain, fatigue, nausea, sadness, anxiety, insomnia, loss of appetite, feeling of well-being and shortness of breath. The severity of each symptom is evaluated with numerical scores from 0 to 10. The most important rule in evaluating the symptom is that the patient marks the number indicating the severity of the symptom according to his/her own statement. The patient is asked to match the symptoms he/she experiences with a number between 0-10 that he/she thinks best fits him/her. A score of 0 on the scale indicates that there is no symptom, while a score of 10 indicates that the symptom is experienced very severely.
EORTC QLQ-C 30 Quality of Life Scale | At the end of Sessions 16 ( each Session 1 days a week)
  It consists of 30 questions with three subscales: general well-being (questions 29, 30), functional difficulties (questions 1-7, 20-27) and symptom control (questions 8-19 and 28). The first 28 items in the scale are four-point Likert. Not at all: 1, A little: 2, Quite a bit: 3, A lot: 4 points. These items are questions regarding symptoms and functional domain. Low scores on these items indicate high quality of life, while high scores indicate low quality of life.
Brief Psychological Resilience Scale | At the end of Sessions 16 ( each Session 1 days a week)
  It is a 5-point Likert type, 6-item, self-report measurement tool. It has an answer key of "Not at all appropriate" (1), "Not Applicable" (2), "Somewhat Appropriate" (3), "Appropriate" (4), "Completely Appropriate". Items 2, 4, and 6 in the scale are reverse coded. High scores obtained after translating the reverse coded items indicate a high level of psychological resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No